CLINICAL TRIAL: NCT01643967
Title: Clinical Trial, Open, Phase III, Multicenter, Randomized to Evaluate the Efficacy and Safety of the Use of Ozone Released by Philozon Medplus Device Versus Conventional Therapy in Treating Patients With Diabetic Foot.
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of the Use of Ozone Versus Sunflower Oil in Treating Diabetic Foot
Acronym: PHIOZO0110
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philozon Geradores de Ozonio LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHI-OZO-01-10
Record Dates: First submitted 2012-06-29; First posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus
Keywords: Ozone; Sunflower oil; diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sunflower Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ozone therapy (Experimental): The research subject will receive topical and rectal insufflation of ozone three times a week on alternate days for two months or at least 12 sessions.
  Interventions: Other: sunflower oil
- sunflower oil (Active Comparator): The research subjects allocated to this treatment arm will receive Sunflower Oil supplied by Philozon. Sunflower oil should be applied once daily for 60 days, it immediately after cleansing site where the lesion is present.
  Other Names:
  Sunflower oil
  Interventions: Other: Ozone Therapy

INTERVENTIONS:
Other: sunflower oil — The research subjects allocated to this treatment arm will receive Sunflower Oil supplied by Philozon. Sunflower oil should be applied once daily for 60 days, it immediately after cleansing site where the lesion is present.
  Arms: Ozone therapy
Other: Ozone Therapy — The research subject will receive topical and rectal insufflation of ozone three times a week on alternate days for two months or at least 12 sessions.
  Other Names: Philozon, MedPlus, Ozone Therapy
  Arms: sunflower oil

SUMMARY:
This is a open, phase III, multicenter, prospective, comparative, controlled, randomized clinical trial to evaluate the efficacy and safety of the use of ozone released by Philozon Medplus device versus conventional therapy in treating patients with diabetic foot.

DETAILED DESCRIPTION:
* Clinical trial, open, phase III, multicenter, prospective, comparative, controlled, randomized to evaluate the efficacy and safety of the use of ozone released by Philozon Medplus device versus conventional therapy in treating patients with diabetic foot.
* Primary Objective: evaluate the efficacy and safety of ozone released by the device Philozon Medplus in the treatment of patients with diabetic foot.
* Secondary objective: evaluate ozone analyzer by environmental ozone Philozon Medplus released by the device in the clinical setting after using the device for rectal insufflation in a patient with diabetic foot.
* Study population: Patients of both sexes, consisting of 100 patients over 18 years, patients with diabetic foot.
* Treatment: 50 patients receive ozone therapy (topical and rectal insufflation of ozone). 50 patients will receive conventional treatment (Sunflower Oil).

ELIGIBILITY:
Inclusion Criteria:

* Consent form signed;
* Patients with Diabetes Mellitus Type I or Type II trophic lesions presenting in the lower limbs;
* Injury whose largest diameter is less than 5 cm;
* Patients of both sexes, aged above 18 years;
* Heart rate 60 to 100 bpm.

Exclusion Criteria:

* Presence of severe septic conditions;
* IMC > 30;
* Presence of Lymphedema;
* Presence of trophic lesions in the lower limbs: exudative, traumatic and parasitic;
* Trophic lesions caused by venous disease requiring treatment;
* Hepatic or renal dysfunction;
* History of alcohol abuse and drugs in the last 6 months;
* Laboratory parameters:
* hemoglobin < 10 g/dl;
* Glycated hemoglobin > 9%;
* Diagnosis of hyperthyroidism (TSH < 0.50 μUI/mL, free T4 > 1.80 ng/dL);
* Deficit of Glucose 6 Phosphate Dehydrogenase (G6PD) > 20%;
* Use of immunosuppressive drugs or anticonvulsants;
* Pregnant woman or lactating;
* Any significant medical condition which in the opinion of the Investigator may bring risks to the patient;
* Known hypersensitivity to drugs and/or treatments to be used in the study;
* Inability to compliance with the protocol;
* Participation in another clinical trial for less than 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy and safety of ozone released by the device Philozon Medplus in the treatment of patients with diabetic foot. | 65 days
  Evaluate the efficacy and safety of the release of ozone Medplus Philozon device in the treatment of patients with diabetic foot, through the clinical evaluation by the investigator based on the time needed for healing and decreasing the larger diameter of the lesion to be accompanied by image (photo), which register the size of the lesion in centimeters with a ruler.

SECONDARY OUTCOMES:
Evaluate the release of ozone in the environment by equipment MEdplus after insufflation rectal in patients with diabetic foot. | 65 days
  Evaluate using ozone analyzer environmental ozone released by the device Philozon Medplus in the clinical setting after using the device for rectal insufflation in a patient with diabetic foot.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz L Pfluck, Investigator, Principal Investigator — Pronto Socorro de Fraturas; Marcelo C Burihan, Investigator, Principal Investigator — Hospital Santa Marcelina; Renato t Santos, Investigator, Principal Investigator — Associação Hospitalar Beneficente São Vicente de Paulo
Locations (1):
- Associação Hospitalar Beneficente São Vicente de Paulo, Passo Fundo, Rio Grande do Sul, Brazil